CLINICAL TRIAL: NCT07175129
Title: Transverse Tibial Bone Transport in "No Option" Patients With Chronic Limb-Threatening Ischemia: A Pilot Study
Brief Title: Transverse Tibial Transport for Chronic Limb-Threatening Ischemia (CLTI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Mehdi Shishehbor, MD, President, University Hospitals Harrington Heart and Vascular Institute, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY20250771
Record Dates: First submitted 2025-09-14; First posted 2025-09-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Limb Threatening Ischemia
Keywords: peripheral artery disease; Diabetic Foot
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transverse Tibial Bone Transport Patients (Experimental): Patients in this arm will undergo transverse tibial bone transport
  Interventions: Procedure: Transverse Tibial Bone Transport; Device: TrueLok Elevate

INTERVENTIONS:
Procedure: Transverse Tibial Bone Transport — Tibial tibial bone transport is a novel surgical procedure that involves the gradual movement of a bone segment in order to improve perfusion and tissue healing.
Device: TrueLok Elevate — This device is used to move the bone segment as a part of the tibial bone transport surgery.

SUMMARY:
Chronic limb-threatening ischemia (CLTI) is a serious condition that happens when blood flow to the legs or feet is severely reduced. This can lead to constant pain, wounds that don't heal, infections, and in some cases, the need for amputation.

Some people with CLTI have such severe artery disease that doctors are unable to restore blood flow using standard treatments like surgery or stents. For these patients, major amputation may be the only remaining option.

This study aims to test a new surgical technique called transverse tibial bone transport, which has been shown in some previous small studies to help improve blood flow and promote healing of wounds in the legs and feet. These early studies suggest that the procedure may help wounds heal better and reduce the need for amputation in people with severe circulation problems. This research will help us learn more about how safe and effective this technique is for patients who have no other treatment options other than amputation.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years and under 95 years
* History of diabetes mellitus with stable glycemic control (HbA1C<10)
* Clinical diagnosis of chronic limb-threatening ischemia
* Stable Rutherford Classification 5 or 6 ischemic ulcer on foot
* Subjects who are determined by an independent multidisciplinary team of surgical and endovascular experts to have no feasible conventional distal bypass surgical or endovascular therapy for limb salvage.
* Subjects who are enrolled in an appropriate wound care network and have a sufficient support system to ensure compliance with medication regimens and follow-up study visits.
* Subjects who are willing and able to provide informed consent

Exclusion Criteria:

* Frailty or severe comorbidities including significantly reduced cardiac, hepatic, renal and respiratory insufficiency making the subject not fit for surgery
* Active malignancy or immunodeficiency disorder
* Previous major amputation of the target limb or presence of a wound requiring a free flap
* Life expectancy less than 12 months
* Active infection at the time of the index procedure
* Any significant concurrent medical, psychological, or social condition that, in the opinion of the investigator, may substantially interfere with the subject's optimal participation in the study.
* Pregnancy at the time of enrolment
* The subject participating in another investigational drug or device study that has not completed its primary endpoint or clinically interferes with the endpoints of this study.
* The subject is unwilling or unable to comply with any protocol or follow-up requirements.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients avoiding major amputation | Up to 6 months post surgery
  major amputation refers to the surgical removal of a limb anywhere above the ankle joint
Percentage of patients achieving complete wound healing as measured by the direct wound observation | Up to 6 months post surgery
Percentage of patients achieving a decrease in the Rutherford classification measured by direct observation | Up to 6 months post surgery
  The Rutherford wound classification is an observational technique to assess the severity of peripheral artery disease of the lower limb on a scale of 0 being asymptomatic to 6 being major tissue loss.
Changes in lower extremity arterial perfusion measured by ankle-brachial index and toe-brachial index | 1 month, 3 months, and 6 months post surgery
  The Ankle-Brachial Index (ABI) and Toe-Brachial Index (TBI) are noninvasive measures of lower-extremity arterial perfusion, calculated as the ratio of the highest systolic blood pressure at the ankle or great toe, respectively, to the highest systolic blood pressure at the brachial artery. Lower ABI and TBI values on indicate greater arterial obstruction.

SECONDARY OUTCOMES:
Changes in pain measured by the Visual Analog Scale | 1 week, 2 weeks, 1 month, 2 months, 3 months, and 6 months post surgery
  The Visual Analogue Scale (VAS) is a simple tool used to measure the intensity of pain. It typically consists of a 100 mm horizontal line anchored by two extremes, such as "No pain" on the left and "Worst imaginable pain" on the right.
  Participants mark a point along the line that best represents their experience, and the distance from the "no pain" end to the mark is measured in millimeters to produce a score from 0 to 100.
Changes in lower extremity neuropathy measured by Semmes-Weinstein Monofilament Test | 1 week, 2 weeks, 1 month, 2 months, 3 months, and 6 months post surgery
  The Semmes-Weinstein Monofilament Test is a standardized assessment of light touch and protective sensation using calibrated nylon filaments, with inability to perceive the 10-gram (5.07) monofilament at specified sites indicating loss of protective sensation.
Changes in quality of life measured by the Short Form-36 (SF-36) scores | 1 month, 2 months, 3 months, and 6 months post surgery
  The Short Form-36 (SF-36) Health Survey is a validated 36-item questionnaire assessing eight domains of health-related quality of life, with scores for each domain ranging from 0 to 100, where higher scores indicate better perceived health status.
Percentage of patients experiencing adverse outcomes | Up to 6 months post surgery
  All adverse outcomes and complications directly attributable to the transverse tibial bone transport procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang AA, Park N, Gazes MI, Samchukov M, Frumberg DB. Transverse tibial bone transport for non-healing heel wound: A case report. Int J Surg Case Rep. 2024 Nov;124:110400. doi: 10.1016/j.ijscr.2024.110400. Epub 2024 Oct 2. PMID 39369454
- [Background] Wen R, Cheng X, Cao H, Zhang L, Luo F, Shang W. Transverse Tibial Bone Transfer in the Treatment of Diabetes Foot Ulcer: A Pilot Study. Diabetes Metab Syndr Obes. 2023 Jul 3;16:2005-2012. doi: 10.2147/DMSO.S413884. eCollection 2023. PMID 37427081
- [Background] Yu L, Zhang D, Yin Y, Li X, Bai C, Zhou Q, Liu X, Tian X, Xu D, Yu X, Zhao S, Hu R, Guo F, Yang Y, Ren Y, Chen G, Zeng J, Feng J. Tibial cortex transverse transport surgery improves wound healing in patients with severe type 2 DFUs by activating a systemic immune response: a cross-sectional study. Int J Surg. 2025 Jan 1;111(1):257-272. doi: 10.1097/JS9.0000000000001897. PMID 38954658
- [Background] Zuo Q, Gao F, Song H, Zhou J. Application of Ilizarov transverse tibial bone transport and microcirculation reconstruction in the treatment of chronic ischemic diseases in lower limbs. Exp Ther Med. 2018 Aug;16(2):1355-1359. doi: 10.3892/etm.2018.6321. Epub 2018 Jun 18. PMID 30116386
- [Background] Ou S, Xu C, Yang Y, Chen Y, Li W, Lu H, Li G, Sun H, Qi Y. Transverse Tibial Bone Transport Enhances Distraction Osteogenesis and Vascularization in the Treatment of Diabetic Foot. Orthop Surg. 2022 Sep;14(9):2170-2179. doi: 10.1111/os.13416. Epub 2022 Aug 10. PMID 35946439
- [Background] Hu XX, Xiu ZZ, Li GC, Zhang JY, Shu LJ, Chen Z, Li H, Zou QF, Zhou Q. Effectiveness of transverse tibial bone transport in treatment of diabetic foot ulcer: A systematic review and meta-analysis. Front Endocrinol (Lausanne). 2023 Jan 4;13:1095361. doi: 10.3389/fendo.2022.1095361. eCollection 2022. PMID 36686461
- [Background] Liu J, Yao X, Xu Z, Wu Y, Pei F, Zhang L, Li M, Shi M, Du X, Zhao H. Modified tibial cortex transverse transport for diabetic foot ulcers with Wagner grade >/= II: a study of 98 patients. Front Endocrinol (Lausanne). 2024 Jan 22;15:1334414. doi: 10.3389/fendo.2024.1334414. eCollection 2024. PMID 38318295